CLINICAL TRIAL: NCT02322190
Title: Biomarkers in Acute Graft-Versus-Host Disease (GVHD) and Extracorporeal Photopheresis Added to Investigator Chosen Therapies of Steroid Refractory Acute GVHD
Brief Title: Biomarkers in Acute Graft-Versus-Host Disease and Extracorporeal Photopheresis Added to Investigator Chosen Therapies of Steroid Refractory Acute GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow/insufficient accrual and Principal Investigator left the NIH
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Gress, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150039; 15-C-0039
Record Dates: First submitted 2014-12-20; First posted 2014-12-23 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Chronic Graft vs. Host Disease; Graft vs Host Disease; Graft-Versus-Host Disease
Keywords: Steroid Failure; Immunomodulation; Corticosteroid Therapy
MeSH Terms: conditions — Graft vs Host Disease | interventions — Photopheresis; Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Investigator chosen second line therapy (No Intervention): Investigator chosen second line therapy
- Second line therapy + Extracorporeal Photopheresis (Experimental): Second line therapy in addition to Extracorporeal Photopheresis (ECP)
  Interventions: Procedure: Extracorporeal Photopheresis (ECP); Drug: Methoxsalen

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis (ECP) — Twice weekly for 1 month or Twice every other week for 2 months or Twice during one week per month for 4 months for a total of up to 7 months of treatment.
  Other Names: Extracorporeal Photopheresis
  Arms: Second line therapy + Extracorporeal Photopheresis
Drug: Methoxsalen — Sterile solution used in conjunction with photopheresis procedure.
  Other Names: Oxsoralen-Ultra
  Arms: Second line therapy + Extracorporeal Photopheresis

SUMMARY:
Background:

- Some allogeneic stem cell transplant recipients get acute graft-versus-host disease (GVHD). They always get steroids as the first treatment, but this may not work. Those people where steroids are not enough may benefit from a treatment called extracorporeal photopheresis (ECP). ECP exposes white blood cells to ultraviolet light outside the body. Researchers want to study how certain markers in the blood predict the severity and outcome of acute GVHD and how ECP treatments work for people with acute GVHD. They will also study how these markers in the blood may help predict who should get ECP and its effects on the immune system.

Objectives:

- To learn more about treatments for acute GVHD after allogeneic stem cell transplantation.

Eligibility:

- Adults with acute GVHD enrolled in an National Cancer Institute (NCI) allogeneic transplantation protocol.

Design:

* Transplant physicians will confirm participant eligibility.
* Participants will receive treatment with steroids for their acute GVHD as prescribed by their transplant physician. This will continue while they are enrolled on this study.
* If steroids work in treating their acute GVHD, then every 28 days for 6 months, participants will have:
* a physical exam.
* blood tests.
* If steroids do not work, participants will get additional treatments as prescribed by their transplant physician who may choose to use ECP as a part of this additional treatment. For ECP, blood is removed through an intravenous (IV) catheter. A machine separates the white blood cells from the other blood parts. Those cells are treated with methoxsalen and exposed to ultraviolet light. Then they are returned to the participant through their IV.
* Participants who get ECP will over at least 6 months have:
* veins researched. They may have a catheter placed in a larger vein in the chest or groin.
* multiple blood tests.
* multiple pregnancy tests (if needed).
* multiple ECP procedures.
* At the end of ECP treatment and 6 months after ECP, participants will have additional physical exams and blood tests.

DETAILED DESCRIPTION:
Background:

* Acute graft versus host disease (GVHD) remains a difficult to manage complication of allogeneic hematopoietic stem cell transplantation causing significant morbidity and mortality.
* Biomarkers have recently been described in acute GVHD that have the potential to better predict onset, severity, steroid failure, and non-relapse mortality.
* First line treatment of acute GVHD with high dose corticosteroids will fail in approximately 30% of patients and is associated with significant steroid related complications.
* No second line treatment of acute GVHD after a failure of steroids has been established as a standard approach.
* Choice of second line therapy for acute GVHD is currently based primarily on physician familiarity, existing toxicities, and patient's ability to tolerate new potential toxicities.
* Extracorporeal photopheresis (ECP) is an attractive therapy to combine with other therapies for steroid refractory disease due to a unique mechanism of action involving immunomodulation as well as an extremely low rate of reported side effects and complications.
* Biomarkers may also prove useful in predicting the success or failure of specific treatments for steroid refractory disease, including those combined with ECP.
* This study will allow for collection of biomarker data in patients undergoing allogeneic transplantation on National Cancer Institute (NCI) protocols, including those who develop acute GVHD and investigate their role in predicting outcomes in initial corticosteroid therapy as well as in currently used treatments in the management of patients with steroid refractory acute GVHD with or without the addition of ECP.

Objective:

-To study biomarkers in patients undergoing allogeneic transplantation, with acute GVHD including their ability to predict steroid refractoriness and predict outcome of investigator chosen second line therapies with and without Extracorporeal Photopheresis (ECP).

Eligibility:

- Adult patients on an NCI allogeneic transplantation protocol.

Design:

* Non-randomized, single institution study.
* Research blood for biomarkers will be collected on all patients enrolled.
* ECP will be offered as an addition to investigator chosen treatments in patients who develop steroid refractory acute GVHD.
* The study will enroll a total of up to 450 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to18 years.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Subject must be also enrolled on an National Cancer Institute (NCI) allogeneic transplant protocol.
* Patients must agree to practice effective contraception (both male and female subjects, if the risk of conception exists)The effects of Extracorporeal Photopheresis (ECP) on the developing human fetus are unknown. For this reason and as well as other Methoxsalen used in this trial is in a class of agents that is known to be teratogenic, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for 4 months after the completion of study treatment. Should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform her treating physician immediately.

EXCLUSION CRITERIA:

* Any physical or mental condition that, in the opinion of the principal Investigator (PI), would cause the risk/benefit ratio of participation to be unacceptable.
* Inclusion of ECP in the treatment of any patient is contraindicated by any of the following:
* Unstable hemodynamics requiring vasopressors or other support measures not amenable to or medically appropriate for continuation during the procedure.
* Uncontrolled infection.
* Inability to maintain acceptable venous access.
* Uncontrolled or uncorrectable coagulopathy.
* Pregnant women are excluded from ECP because methoxsalen, an agent utilized for the study procedure, may cause fetal harm. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with methoxsalen, breastfeeding should be discontinued if the mother is treated with methoxsalen. Pregnancy will be evaluated prior to initiation of ECP.
* History of allergic or idiosyncratic/hypersensitivity reactions to 8- methoxypsoralen/psoralen compounds.
* History of a light-sensitive cutaneous disease
* Subjects with aphakia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-12-20 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Gress, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were entered in to the Second Line Therapy + Extracorporeal Photopheresis group.
Groups:
- Investigator Chosen Second Line Therapy: Investigator chosen second line therapy is determined on an individual basis based on standard care and actual site of Graft -versus-Host Disease (GVHD). The frequency or duration of therapy is based on Principal Investigator (PI) discretion.
- Second Line Therapy + Extracorporeal Photopheresis: Second line therapy in addition to Extracorporeal Photopheresis (ECP)
  Extracorporeal Photopheresis (ECP): Twice weekly for 1 month or Twice every other week for 2 months or Twice during one week per month for 4 months for a total of up to 7 months of treatment
  Methoxsalen: Used in conjunction with photopheresis procedure
Period: Overall Study
Arm/Group | Investigator Chosen Second Line Therapy | Second Line Therapy + Extracorporeal Photopheresis
Started | 5 | 0
Completed | 4 | 0
Not Completed | 1 | 0
Not completed — Death on study | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Investigator Chosen Second Line Therapy
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.62 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biomarkers (Serum TIM3, IL-6, Reg-3-a, ST2, LPS-BP, Nitrate, TNFR1, IL-2Ra, CXCL10, and HGF) Present in Blood and/or Tissue Who Were Steroid Refractory After ECP Treatment
Description: In an effort to determine steroid refractoriness after Extracorporeal Photopheresis (ECP) treatment, tissue and blood obtained from participants was examined to see if biomarkers (i.e., Serum T cell immunoglobulin and mucin domain-containing protein 3 (TIM3), ST2, Nitrate, Interleukin-6 (IL-6), regenerating family member 3 alpha (Reg-3-a), lipopolysaccharide binging protein (LPS-BP), tumor necrosis factor receptor 1 (TNFR1), interleukin-2 receptor alpha chain (IL-2Ra), CXC motif chemokine 10 (CXCL10), hepatocyte growth factor (HGF)) were present.
Time Frame: 14 Days
Population: No data was collected for this outcome measure and it not done because biomarker studies require large patient numbers to analyze data. Only five participants were enrolled in this study. With early termination, there are no biomarker data to report.
Arm/Group | Investigator Chosen Second Line Therapy
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Steroid Refractory Disease Who Had Improvement and/or Resolution of Graft-versus-host Disease (GVHD) Associated Symptoms
Description: GVHD associated symptoms was assessed by the American Society for Bone Marrow Transplantation consensus statement. Complete Response (CR) is no residual organ specific symptoms or findings. Very Good Partial Response (VGPR) is Skin: An active erythematous rash involving < 25% of the body surface area; Liver: Persistent low-level hyperbilirubinemia, and/or Gut: Gastrointestinal function and water resorption in the colon are approaching normal. Partial Response (PR) is any improvement over baseline symptoms. Progressive disease (PD) is stable or worsening organ specific findings requiring change of therapy.
Time Frame: 7 months
Measure: Count of Participants; unit: Participants
Arm/Group | Investigator Chosen Second Line Therapy
Number analyzed (Participants) | 5
Participants | 2

3. Secondary Outcome: Days to Overall Survival
Description: Overall survival is defined as the time from study entry to end of observations/off study.
Time Frame: time from study entry to end of observations/off study, up to a year
Measure: Median (Full Range); unit: Days
Arm/Group | Investigator Chosen Second Line Therapy
Number analyzed (Participants) | 5
Days | 180 [117 to 318]

4. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 8 months and 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Investigator Chosen Second Line Therapy
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 8 months and 6 days.
Description: No participants were entered in to the Second Line Therapy + Extracorporeal Photopheresis group.
Arm/Group | Investigator Chosen Second Line Therapy | Second Line Therapy + Extracorporeal Photopheresis
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigator Chosen Second Line Therapy (N=5) | Second Line Therapy + Extracorporeal Photopheresis (N=0)
Death (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02322190/Prot_SAP_000.pdf
  • Informed Consent Form (2014-11-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT02322190/ICF_001.pdf